CLINICAL TRIAL: NCT01712243
Title: Toileting at Night in Older Adults: Light to Maximize Vision, Minimize Insomnia
Brief Title: Light to Maximize Vision, Minimize Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Assistant Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1I21RX000773-01A2 (NIH)
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Postural Balance
MeSH Terms: interventions — Light

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dim light (Active Comparator): 15 minutes of very dim (<1 lux) light during the night
  Interventions: Other: Light
- Room light (Active Comparator): 15 minutes of normal room light (~100 lux) during the night
  Interventions: Other: Light
- Colored light (Experimental): 15 minutes of colored light during the night
  Interventions: Other: Light

INTERVENTIONS:
Other: Light

SUMMARY:
The purpose of this study is to determine whether specific wavelengths of light at night can be used to improve mobile balance while simultaneously not increasing alertness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-85
* At least 20/200 corrected visual acuity
* Greater than 20° visual field with no lower visual field loss
* Stable health
* Male or female
* Normal color vision
* Normal hearing

Exclusion Criteria:

* Extreme chronotype
* Sleep disorders
* Dementia
* Smoker
* Depression
* Alcohol abuse
* Use of illegal drugs
* Use of sleep/wake altering drugs on an acute or as needed basis (including nutraceuticals, antihistamines)
* Use of light sensitizing drugs
* Self-reported history of nocturia (>3 times per night)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mobile balance | 15 minutes
  Mobile balance as determined using a GaitRite walkway
Alertness | 15 minutes
  Alertness as determined by electroencephalographic power density

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States